CLINICAL TRIAL: NCT04763044
Title: Evaluation of the Fluoride Dose Response of MFP Dentifrice Using In Situ Caries Model
Brief Title: Evaluation of the Fluoride Dose Response Using In Situ Caries Model
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2020154
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Fifth leg of the study will not be randomized, participants will remain blinded but all will use the same product.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Period 1 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 2 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 3 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 4 (Other): 0 ppm F (placebo, negative control), 250 ppm F as MFP (dose-response control), 1100 ppm F as MFP (reference), 2800 ppm F as MFP (dose-response control)
  Interventions: Drug: 0 ppm F; Drug: 250 ppm F as MFP; Drug: 1100 ppm as MFP; Drug: 2800 ppm F as MFP
- Period 5 (Other): 1100 ppm SnF2 toothpaste only
  Interventions: Drug: 1100 ppm SnF2

INTERVENTIONS:
Drug: 0 ppm F — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
  Arms: Period 1; Period 2; Period 3; Period 4
Drug: 250 ppm F as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
  Arms: Period 1; Period 2; Period 3; Period 4
Drug: 1100 ppm as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
  Arms: Period 1; Period 2; Period 3; Period 4
Drug: 2800 ppm F as MFP — Each subject will be randomly assigned to this treatment during one of the four periods for this crossover study.
  Arms: Period 1; Period 2; Period 3; Period 4
Drug: 1100 ppm SnF2 — Each subject will be assigned to this treatment during the fifth period for this crossover study.
  Arms: Period 5

SUMMARY:
The purpose of this study is to evaluate the fluoride dose response of different dentifrice fluoride concentrations - 0, 250, 1100 and 2800 ppm fluoride as sodium monofluorophosphate (MFP) and a fifth leg of 1100 ppm Stannous Fluoride (SnF2) using an in situ caries model.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 85 years of age;
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be in general good health as determined by the Investigator based on a review of the health history/update for participation in the trial;
* Be wearing a removable mandibular partial denture with sufficient room in one posterior buccal flange area to accommodate two 4 mm round enamel specimens and room on the same side to accommodate two 4 mm round specimens in the buccal surface of two posterior denture teeth;
* Be willing and capable of wearing their removable partial denture 24 hours a day for four (4), three-week treatment periods;
* Be willing to allow study personnel to drill specimen sites (as described in #iv) in their mandibular partial denture;
* Be in good medical and dental health with no active caries or periodontal disease (NOTE: subjects presenting at screening with caries may continue in the study if their carious lesions are restored prior to beginning treatment 1);
* Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate ≥ 0.2 mL/min; gum base stimulated whole saliva flow rate ≥ 0.8 mL/min).

Exclusion Criteria:

* Currently being pregnant, intending to become pregnant during the study period, or breast feeding;
* Currently having any medical condition that could be expected to interfere with the subject's safety during the study period;
* Currently taking antibiotics or having taken antibiotics in the two weeks prior to beginning treatment 1;
* Having participated in another clinical study or receipt of an investigational drug within 30 days of beginning treatment 1; or
* Taking fluoride supplements, required to use a fluoride mouth rinse, or have received a professional fluoride treatment in the two weeks preceding specimen placement;
* Currently taking or have ever taken bisphosphonate drugs (e.g., Fosamax, Actonel and Boniva) for the treatment of osteoporosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Health Research Institute, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2: This was a 4-way crossover design study. All participants were randomized to receive the following interventions in this order: 0, 250, 1100 and 2800 ppm fluoride as sodium monofluorophosphate (MFP) using an in situ caries model. Participants were additionally invited to participate in a fifth leg which contained 1100 ppm SnF2.
- 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2: This was a 4-way crossover design study. All participants were randomized to receive the following interventions in this order: 250, 2800, 0, and 1100 ppm fluoride as sodium monofluorophosphate (MFP) using an in situ caries model. Participants were additionally invited to participate in a fifth leg which contained 1100 ppm SnF2.
- 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2: This was a 4-way crossover design study. All participants were randomized to receive the following interventions in this order: 1100, 0, 2800 and 250 ppm fluoride as sodium monofluorophosphate (MFP) using an in situ caries model. Participants were additionally invited to participate in a fifth leg which contained 1100 ppm SnF2.
- 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2: This was a 4-way crossover design study. All participants were randomized to receive the following interventions in this order: 2800, 1100, 250 and 0 ppm fluoride as sodium monofluorophosphate (MFP) using an in situ caries model. Participants were additionally invited to participate in a fifth leg which contained 1100 ppm SnF2.
Period: Period 1
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2
Started | 3 | 4 | 4 | 4
Completed | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2
Started | 3 | 4 | 4 | 3
Completed | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2
Started | 3 | 4 | 4 | 3
Completed | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2
Started | 3 | 3 | 4 | 3
Completed | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2
Started | 3 | 3 | 4 | 3
Completed | 2 | 3 | 4 | 3
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2: This was a 4-way crossover design study. All participants were randomized to receive the following interventions in this order: 250, 2800, 0 and 1100 ppm fluoride as sodium monofluorophosphate (MFP) using an in situ caries model. Participants were additionally invited to participate in a fifth leg which contained 1100 ppm SnF2.
- Total: Total of all reporting groups
Arm/Group | 0 Ppm MFP, 250 Ppm MFP, 1100 Ppm MFP, 2800 Ppm MFP, 1100 Ppm SnF2 | 250 Ppm MFP, 2800 Ppm MFP, 0 Ppm MFP, 1100 Ppm MFP, 1100 Ppm SnF2 | 1100 Ppm MFP, 0 Ppm MFP, 2800 Ppm MFP, 250 Ppm MFP, 1100 Ppm SnF2 | 2800 Ppm MFP, 1100 Ppm MFP, 250 Ppm MFP, 0 Ppm MFP, 1100 Ppm SnF2 | Total
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.33) | 72.5 (4.51) | 69.7 (9.50) | 76.3 (9.32) | 72.2 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 2 | 9
  Male | 2 | 2 | 0 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 4 | 9
  White | 2 | 2 | 1 | 0 | 5
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Enamel Fluoride Uptake (EFU)
Description: The EFU test will evaluate the level of fluoride in partially demineralized enamel specimens via the microdrill enamel biopsy technique by [Sakkab et al., 1984]. The calculated scores will be measured in μg F/cm2.
Time Frame: Evaluations will occur after 21 days of product use
Measure: Mean (Standard Error); unit: μg F/cm^2
Groups:
- 0 Ppm F (Placebo, Negative Control): Each subject was randomly assigned to 0 ppm F dentifrice during one of the four periods for this crossover study.
- 250 Ppm F as MFP (Dose-response Control): Each subject was randomly assigned to 250 ppm F dentifrice during one of the four periods for this crossover study.
- 1100 Ppm F as MFP (Reference): Each subject was randomly assigned to 1100 ppm F dentifrice during one of the four periods for this crossover study.
- 2800 Ppm F as MFP (Dose-response Control): Each subject was randomly assigned to 2800 ppm F dentifrice during one of the four periods for this crossover study.
- 1100 Ppm SnF2: Each subject was assigned to 1100 ppm SnF2 dentifrice during the fifth period for this study.
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 12
μg F/cm^2 | 2.28 (0.709) | 4.51 (0.709) | 8.78 (0.736) | 14.05 (0.709) | 7.43 (0.423)

2. Secondary Outcome: Enamel Fluoride Uptake (EFU)
Description: as for outcome 1
Time Frame: Evaluations will occur after 7 days of product use
Measure: Mean (Standard Error); unit: μg F/cm^2
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 13
μg F/cm^2 | 3.13 (0.881) | 5.20 (0.882) | 8.20 (0.916) | 13.52 (0.850) | 9.11 (0.670)

3. Secondary Outcome: Percent Surface Microhardness (SMH)
Description: The SMH test will evaluate changes in the mineral status of partially demineralized enamel specimens through use of a Wilson 2100 Hardness Tester. These scores will be calculated as a percent.
Time Frame: Evaluations will occur after 7 days of product use
Measure: Mean (Standard Error); unit: Percent SMH Recovery
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 13
Percent SMH Recovery | 15.92 (3.259) | 22.50 (3.264) | 22.42 (3.360) | 35.61 (3.160) | 26.32 (4.605)

4. Secondary Outcome: Enamel Fluoride Uptake (EFU)
Description: as for outcome 1
Time Frame: Evaluations will occur after 14 days of product use
Measure: Mean (Standard Error); unit: μg F/cm^2
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 13
μg F/cm^2 | 3.86 (1.141) | 7.23 (1.141) | 11.53 (1.185) | 18.92 (1.141) | 12.65 (1.215)

5. Secondary Outcome: Percent Surface Microhardness (SMH)
Description: as for outcome 3
Time Frame: Evaluations will occur after 14 days of product use
Measure: Mean (Standard Error); unit: Percent SMH Recovery
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 13
Percent SMH Recovery | 10.49 (4.258) | 18.62 (4.258) | 24.76 (4.369) | 38.08 (4.258) | 28.28 (4.562)

6. Secondary Outcome: Percent Surface Microhardness (SMH)
Description: as for outcome 3
Time Frame: Evaluations will occur after 21 days of product use
Measure: Mean (Standard Error); unit: Percent SMH Recovery
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
Number analyzed (Participants) | 14 | 14 | 13 | 14 | 12
Percent SMH Recovery | 4.76 (4.921) | 11.14 (4.921) | 17.51 (5.068) | 33.38 (4.921) | 17.91 (3.108)

ADVERSE EVENTS:
Time Frame: Each participant was monitored throughout the whole study, up to 4 months.
Arm/Group | 0 Ppm F (Placebo, Negative Control) | 250 Ppm F as MFP (Dose-response Control) | 1100 Ppm F as MFP (Reference) | 2800 Ppm F as MFP (Dose-response Control) | 1100 Ppm SnF2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 3/14 | 2/14 | 2/13 | 5/14 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0 Ppm F (Placebo, Negative Control) (N=14) | 250 Ppm F as MFP (Dose-response Control) (N=14) | 1100 Ppm F as MFP (Reference) (N=13) | 2800 Ppm F as MFP (Dose-response Control) (N=14) | 1100 Ppm SnF2 (N=13)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Irritation Mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Edentulous Ridge Erythmea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vaginitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Tooth Broken (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Neck Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Renal Kidney Tumor (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Irritation Gum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Irritation Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI should disclose plans to sponsor prior to public release.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT04763044/Prot_SAP_000.pdf